CLINICAL TRIAL: NCT04699955
Title: Longitudinal Use of Protective Behavioral Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SBE-17-13260
Record Dates: First submitted 2020-05-22; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Alcohol Use, Unspecified
Keywords: Deviance Regulation Theory; Alcohol Use; Alcohol Consequences; Protective Behavioral Strategies; College Freshman
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to 1 of 3 parallel conditions. After assignment, they received a brief intervention and were then followed for the next 12 months.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Assessment only Control (No Intervention): Participants received no intervention content. They provided assessments of past week protective strategy use, alcohol use, and alcohol problems. All assessments were delivered via an online survey.
- Positive Message Condition (Experimental): Participants received information on the positive aspects of individuals that used protective strategies and were encouraged to report why these individuals were viewed so much more positively. They provided assessments of past week protective strategy use, alcohol use, and alcohol problems. All assessments and messaging was delivered via an online survey.
  Interventions: Behavioral: Deviance Regulation Theory
- Negative Message Condition (Experimental): Participants received information on the negative aspects of individuals that did not used protective strategies and were encouraged to report why these individuals were viewed so much more negatively. They provided assessments of past week protective strategy use, alcohol use, and alcohol problems. All assessments and messaging was delivered via an online survey.
  Interventions: Behavioral: Deviance Regulation Theory

INTERVENTIONS:
Behavioral: Deviance Regulation Theory — In the negative message condition, participants received information on the negative aspects of individuals that did not used protective strategies and were encouraged to report why these individuals were viewed so much more negatively. In the positive message condition, participants received information on the positive aspects of individuals that used protective strategies and were encouraged to report why these individuals were viewed so much more positively.
  Arms: Negative Message Condition; Positive Message Condition

SUMMARY:
This study tested a deviance regulation theory intervention in a sample of university freshman. The aims were to (a) increase use of protective behavioral strategies, (b) decrease alcohol use, and (c) decrease alcohol-related consequences.

DETAILED DESCRIPTION:
College student freshmen were invited to participate in a study on the use of alcohol protective behavioral strategies. They were randomly assigned to receive a positive message about individuals that used protective strategies, a negative message about individuals that did not use protective strategies, or an assessment control. They were then followed for the next 12 months. Assessments were completed at weeks 0, 1, 2, 3, 4, 5, 12, 26, and 52.

ELIGIBILITY:
Inclusion Criteria:

* College freshman at UCF
* Endorse alcohol consumption in the past two weeks

Exclusion Criteria:

* Severe mental illness
* Under 18 years of age
* Over 21 years of age
* Unable to speak English fluently

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2019-08-13 (Actual)

PRIMARY OUTCOMES:
Protective Behavioral Strategies- Pre-Intervention | Past three months prior to intervention/study
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past three months.
Protective Behavioral Strategies- Initial intervention (Week 1) | Past week before intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past week.
Protective Behavioral Strategies- Week 2 | Past 1 week measured- 1 week post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past week.
Protective Behavioral Strategies- Week 3 | Past 1 week measured-2 weeks post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past week.
Protective Behavioral Strategies- Week 4 | Past 1 week measured-3 weeks post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past week.
Protective Behavioral Strategies- Week 5 | Past 1 week measured-4 weeks post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past week.
Protective Behavioral Strategies- Week 6 | Past 1 week measured-5 weeks post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past week.
Protective Behavioral Strategies- 3 month follow up | Past 3 months measured- 12 week post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past three months.
Protective Behavioral Strategies- 6 month follow-up | Past 3 months measured- 26 weeks post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past three months.
Protective Behavioral Strategies- 12 month follow-up | Past 3 months measured- 52 weeks post intervention
  Protective behavioral strategies (PBS) are a collection of harm-reduction strategies aimed to decrease alcohol-related consequences when consuming alcohol. The are three broad subtypes of PBS: (1) Manner of Drinking (MD; e.g., avoiding mixing different types of alcohol), (2) Stopping/Limiting Drinking (SLD; e.g., stopping drinking at a predetermined time), and (3) Serious Harm Reduction (SHR; e.g., knowing where your drink is at all times).
  These PBS were assessed in this study using Protective Behavioral Strategies Survey-20 (PBS-20). The PBS-20 consists of 20 statements covering three factors of protective strategies: Manner of Drinking, Stopping/Limiting Drinking, and Serious Harm Reduction. The frequency of PBS use was be reported on a five-point Likert-scale from 'Never' to 'Always'. Participants were asked to record their PBS use from the past three months.

SECONDARY OUTCOMES:
Alcohol-related consequences- Pre-intervention | Past three months prior to intervention/study
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past three months.
Alcohol-related consequences- Initial intervention (Week 1) | Past week before intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past week.
Alcohol-related consequences- Week 2 | Past 1 week measured- 1 week post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past week.
Alcohol-related consequences- Week 3 | Past 1 week measured- 2 week post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past week.
Alcohol-related consequences- Week 4 | Past 1 week measured- 3 week post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past week.
Alcohol-related consequences- Week 5 | Past 1 week measured- 4 week post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past week.
Alcohol-related consequences- Week 6 | Past 1 week measured- 5 week post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past week.
Alcohol-related consequences- 3 month follow up | Past 3 months measured- 12 week post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past three months.
Alcohol-related consequences- 6 month follow-up | Past 3 months measured- 26 weeks post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past three months.
Alcohol-related consequences- 12 month follow-up | Past 3 months measured- 52 weeks post intervention
  Alcohol-related consequences was assessed using the Young Adult Alcohol Consequences Questionnaire (YAACQ), which consists of 48 items assessing eight categories of alcohol-related consequences: Social-Interpersonal, Impaired Control, Self-Perception, Self-Care, Risk Behaviors, Academic/Occupational, Physical Dependence, and Blackout Drinking. Participants recorded alcohol consequences (Yes/No/ I do not wish to respond) from the past three months.
Alcohol use- Pre-intervention | Past three months prior to intervention/study
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure average alcohol consumption and time spent drinking during a typical week over the past three months. The DDQ-M is composed of a free-text grid where individuals report the number of drinks typically consumed for each day of the week for the past three months.
Alcohol use- Initial intervention (Week 1) | Past week before intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure the number of drinks consumed for each day of the past week. Each grid began with Monday and ended with Sunday, as surveys were sent out on Mondays.
Alcohol use- Week 2 | Past 1 week measured- 1 week post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure the number of drinks consumed for each day of the past week. Each grid began with Monday and ended with Sunday, as surveys were sent out on Mondays.
Alcohol use- Week 3 | Past 1 week measured- 2 weeks post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure the number of drinks consumed for each day of the past week. Each grid began with Monday and ended with Sunday, as surveys were sent out on Mondays.
Alcohol use- Week 4 | Past 1 week measured- 3 weeks post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure the number of drinks consumed for each day of the past week. Each grid began with Monday and ended with Sunday, as surveys were sent out on Mondays.
Alcohol use- Week 5 | Past 1 week measured- 4 weeks post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure the number of drinks consumed for each day of the past week. Each grid began with Monday and ended with Sunday, as surveys were sent out on Mondays.
Alcohol use- Week 6 | Past 1 week measured- 5 weeks post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure the number of drinks consumed for each day of the past week. Each grid began with Monday and ended with Sunday, as surveys were sent out on Mondays.
Alcohol use- 3 month follow up | Past 3 months measured- 12 week post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure average alcohol consumption and time spent drinking during a typical week over the past three months. The DDQ-M is composed of a free-text grid where individuals report the number of drinks typically consumed for each day of the week for the past three months.
Alcohol use- 6 month follow up | Past 3 months measured- 24 week post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure average alcohol consumption and time spent drinking during a typical week over the past three months. The DDQ-M is composed of a free-text grid where individuals report the number of drinks typically consumed for each day of the week for the past three months.
Alcohol use- 12 month follow up | Past 3 months measured- 52 week post intervention
  Alcohol use (quantity) was assessed using the Modified Daily Drinking Questionnaire (DDQ-M). The DDQ-M was used to measure average alcohol consumption and time spent drinking during a typical week over the past three months. The DDQ-M is composed of a free-text grid where individuals report the number of drinks typically consumed for each day of the week for the past three months.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be stored at the Open Science Framework
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: At completion of study
URL: https://osf.io/akef9/

REFERENCES:
- [Derived] Leary AV, Dvorak RD, Troop-Gordon W, Blanton H, Peterson R, Kramer MP, De Leon AN, Magri T. Test of a deviance regulation theory intervention among first-year college student drinkers: Differential effects via frequency and quantity norms. Psychol Addict Behav. 2022 Sep;36(6):619-634. doi: 10.1037/adb0000777. Epub 2021 Sep 30. PMID 34591518
- Available data/document: Individual Participant Data Set — https://osf.io/akef9/